CLINICAL TRIAL: NCT02349711
Title: Probiotics (Lactobacillus Gasseri KS-13, Bifidobacterium Bifidum G9-1, Bifidobacterium Longum MM-2) and Health-related Quality of Life in Individuals With Seasonal Allergies
Brief Title: Probiotics and Health-related Quality of Life in Individuals With Seasonal Allergies
Acronym: JEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Wakunaga Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB201400894; Project No. 00120905 (Other: Wakunaga Pharmaceutical Co., Ltd.)
Record Dates: First submitted 2015-01-23; First posted 2015-01-29 (Estimated); Results first posted 2016-08-31 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Healthy
Keywords: probiotic; allergy; immune
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo will be taken as a capsule twice daily for 8 weeks by subjects in the group receiving this supplement (group is unknown, double-blinded).
  Interventions: Dietary Supplement: Placebo
- Probiotic mixture (Experimental): A commercially available probiotic mixture of Lactobacillus gasseri, Bifidobacterium bifidum, and Bifidobacterium longum will be taken as a capsule twice daily for 8 weeks by subjects in the group receiving this supplement (group is unknown, double-blinded).
  Interventions: Dietary Supplement: Probiotic mixture

INTERVENTIONS:
Dietary Supplement: Probiotic mixture — A 350 mg capsule containing a mixture of Lactobacillus gasseri, Bifidobacterium bifidum, and Bifidobacterium longum (1.5 billion cells per capsule prior to expiration) will be taken twice daily for 8 weeks by subjects in the group receiving this supplement (group is unknown, double-blinded). Inactive ingredients include gelatin, potato starch, and silica.
  Other Names: Kyo-Dophilus; Lactobacillus gasseri KS-13; Bifidobacterium bifidum G9-1; Bifidobacterium longum MM-2
  Arms: Probiotic mixture
Dietary Supplement: Placebo — Placebo will be taken as a capsule twice daily for 8 weeks by subjects in the group receiving this supplement (group is unknown, double-blinded). Supplement contains 348.25 mg of potato starch.
  Arms: Placebo

SUMMARY:
In this randomized, double-blind, placebo-controlled study, participants with seasonal allergies will receive a daily probiotic or placebo for 8 weeks. Questionnaires will assess health-related quality of life, stress, physical activity, gastrointestinal symptoms, adverse events, and compliance. In a subset of subjects, stool and blood samples will be collected at baseline and at week 6 of the intervention (estimated to be peak allergy season) to characterize microbial communities and immune function.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be included if they:

* are 18 to 60 years of age (inclusive).
* receive a score of 2 or greater on the Mini Rhinoconjunctivitis Quality of Life Questionnaire.
* are willing and able to complete the Informed Consent Form in English.
* are available for 8 consecutive weeks to participate in this study.
* be willing and able to complete online daily and weekly questionnaires regarding general wellness, bowel function, quality of life, gastrointestinal symptoms, and physical activity.
* are willing and able to maintain their regular level of physical activity and diet for the 8-week study.
* are able to take the study supplement without the aid of another person.
* are willing to discontinue consumption of fermented foods or probiotics (e.g., yogurts with live, active cultures or supplements), or immune-enhancing supplements (e.g., Echinacea or fish oil).
* are willing to provide 2 blood and 2 stool samples (subgroup only).

Exclusion Criteria:

Subjects will be excluded if they:

* do not meet any of the above criteria.
* use allergy medications, including nasal sprays, 5 or more days per week.
* receive allergy shots.
* are currently pregnant or attempting to get pregnant.
* are currently taking any systemic corticosteroids, androgens (such as testosterone), or large doses of anti-inflammatory drugs (i.e., aspirin in doses >600 mg/d) on a regular basis.
* are currently being treated for or have any of the following physician-diagnosed diseases or conditions: HIV/AIDS; immune modulating diseases (autoimmune disease, hepatitis, cancer, etc.); kidney disease; pancreatitis; pulmonary disease; hepatic or biliary disease; or gastrointestinal diseases/conditions such as diverticulitis, ulcerative colitis, Crohn's disease, Celiac disease, short bowel disease, ileostomy, or colostomy, but not including GERD; or have a central venous catheter.
* have received chemotherapy or other immune suppressing therapy within the last year.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 224 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bobbi Langkamp-Henken, PhD, RD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] Dennis-Wall JC, Culpepper T, Nieves C Jr, Rowe CC, Burns AM, Rusch CT, Federico A, Ukhanova M, Waugh S, Mai V, Christman MC, Langkamp-Henken B. Probiotics (Lactobacillus gasseri KS-13, Bifidobacterium bifidum G9-1, and Bifidobacterium longum MM-2) improve rhinoconjunctivitis-specific quality of life in individuals with seasonal allergies: a double-blind, placebo-controlled, randomized trial. Am J Clin Nutr. 2017 Mar;105(3):758-767. doi: 10.3945/ajcn.116.140012. Epub 2017 Feb 22. PMID 28228426

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Gainesville, FL area, including the University of Florida campus. Recruiting began in January of 2015 and took place in facilities within the Food Science and Human Nutrition Department at the University of Florida. Participants were enrolled from 1-20-15 to 3-12-15.
Pre-assignment Details: Before randomization, participants provided anthropometric measurements and demographic information. Out of the 224 participants who consented to participate, only 173 remained at randomization due to the participants no longer being interested or not coming to their study visits to be randomized.
Groups:
- Placebo: Placebo was to be taken as a capsule twice daily for 8 weeks by subjects in the group receiving this supplement (group was unknown, double-blinded). Supplement contains 348.25 mg of potato starch.
- Probiotic Mixture: A 350 mg capsule containing a commercially available probiotic mixture of Lactobacillus gasseri, Bifidobacterium bifidum, and Bifidobacterium longum (1.5 billion cells per capsule prior to expiration) was to be taken as a capsule twice daily for 8 weeks by subjects in the group receiving this supplement (group was unknown, double-blinded). Inactive ingredients included gelatin, potato starch, and silica.
Period: Overall Study
Arm/Group | Placebo | Probiotic Mixture
Started | 87 | 86
Completed | 84 | 84
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Probiotic Mixture | Total
Number analyzed (Participants) | 87 | 86 | 173
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.6 (13.1) | 26.0 (10.8) | 26.8 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 54 | 119
  Male | 22 | 32 | 54

OUTCOME MEASURES:

1. Primary Outcome: Change in Health-related Quality of Life Score From Baseline to the Peak Week of Allergy Season for Probiotic Versus Placebo, as Measured by MiniRQLQ
Description: MiniRQLQ, global score (0=not troubled, 6=extremely troubled; an average of the 14 questions; includes all domains)
Time Frame: up to 8 weeks from date of randomization
Population: Because this was an intent-to-treat study, all data from all randomized participants was considered for analysis. No imputation was done, so missing values excluded a participant from the analysis. While data from a participant may be missing, they were considered to have "completed" the study if they completed all study visits.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Probiotic Mixture
Number analyzed (Participants) | 80 | 81
units on a scale | -0.1946 (0.1386) | -0.6772 (0.1302)

2. Secondary Outcome: Serum Total Immunoglobulin E (IgE)
Description: Serum total immunoglobulin E (IgE) was quantified via ELISA
Time Frame: baseline and week 6
Population: A subgroup of participants who completed the main study (questionnaire data only) also completed an additional portion of the study in which they provided blood and stool samples.
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Probiotic Mixture
Number analyzed (Participants) | 37 | 35
ng/mL
  Baseline | 325.3243243 (51.4187025) | 781.0285714 (103.2435603)
  Week 6 | 352.6111111 (56.5615450) | 843.3428571 (107.3421604)

3. Secondary Outcome: Constipation Symptom Score, Measured by Gastrointestinal Symptom Response Scale (GSRS) Questionnaire
Description: Symptoms included in this score are constipation, hard stools, and feeling of incomplete evacuation reported on a weekly Gastrointestinal Symptom Response Scale (GSRS) questionnaire. Questionnaire asks participants about the previous seven days. Scores range from 1 (no discomfort) to 7 (very severe discomfort); lower scores are more desirable.
Time Frame: weeks 0, 1, 2, 3, 4, 5, 6, 7
Population: Since this outcome had more than two time points, and since all randomized participants provided some weeks of survey data, all participants were included in the analysis (even those that were lost to follow up). The number of values (and thus the number analyzed) by week is also shown.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Probiotic Mixture
Number analyzed (Participants) | 87 | 86
units on a scale
  Week 0: number analyzed (Participants) | 84 | 82
  Week 0 | 1.57 (0.09) | 1.51 (0.08)
  Week 1: number analyzed (Participants) | 83 | 82
  Week 1 | 1.51 (0.08) | 1.49 (0.08)
  Week 2: number analyzed (Participants) | 85 | 83
  Week 2 | 1.59 (0.09) | 1.53 (0.08)
  Week 3: number analyzed (Participants) | 82 | 81
  Week 3 | 1.68 (0.09) | 1.42 (0.07)
  Week 4: number analyzed (Participants) | 77 | 80
  Week 4 | 1.73 (0.11) | 1.41 (0.07)
  Week 5: number analyzed (Participants) | 81 | 81
  Week 5 | 1.61 (0.08) | 1.48 (0.07)
  Week 6: number analyzed (Participants) | 82 | 82
  Week 6 | 1.60 (0.08) | 1.37 (0.06)
  Week 7: number analyzed (Participants) | 82 | 80
  Week 7 | 1.65 (0.08) | 1.31 (0.06)

4. Secondary Outcome: Regulatory T Cells (Tregs)
Description: Regulatory T cells (Tregs) as a percentage of CD4+ T cells, quantified via flow cytometry
Time Frame: baseline and week 6
Population: A subgroup of participants who completed the main study (questionnaire data only) also completed an additional portion of the study in which they provided blood and stool samples. Some samples could not be accurately measured for this outcome, so those samples were excluded from analysis.
Measure: Least Squares Mean (Standard Error); unit: percentage of CD4+ T lymphocytes
Arm/Group | Placebo | Probiotic Mixture
Number analyzed (Participants) | 35 | 35
percentage of CD4+ T lymphocytes
  Baseline | 4.1931 (0.2427) | 4.4146 (0.2533)
  Week 6 | 4.7733 (0.2004) | 4.8626 (0.2007)

ADVERSE EVENTS:
Arm/Group | Placebo | Probiotic Mixture
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/86
Other Adverse Events (participants affected / at risk) | 0/87 | 0/86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall provide the sponsor copies of any proposed publication or presentation at least 30 days in advance of submission to a journal, editor, or other third party to allow sponsor to determine whether patentable subject matter or sponsor's confidential information would be disclosed.